CLINICAL TRIAL: NCT03641027
Title: Physical Activity Before Obesity Surgery
Acronym: PABOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Borås Lasarett (Other); Centrallasarettet i Växjö (Unknown); Karlshamns lasarett (Unknown); Torsby sjukhus (Unknown); Mora sjukhus (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FoU i VGR: 202291
Record Dates: First submitted 2018-08-06; First posted 2018-08-21 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Physical Activity
Keywords: Obesity; Physical Activity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel Assignment A single blind, randomized, controlled, intervention study. Evaluation of the addition of increased physical activity for patients undergoing obesity surgery compared to standard care.
Who Masked: Outcomes Assessor
Masking Description: Assessor will not be aware of which group the patients are included in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Increased physical activity (Experimental): Increased physical activity daily before surgery. Standard care during hospital stay and continued training after discharge.
  Interventions: Other: Increased physical activity
- Standard care (Other): Standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Increased physical activity — Preoperatively
  Individual coaching by a physical therapist to:
  * increase physical activity 30 minutes/day (At least 150 min/week)
  * decrease time spent sitting/lying
  Telephone follow up one week after the intervention starts
  At the hospital
  -Frequent mobilization
  After discharge
  A telephone follow up one week postoperatively with coaching by a physical therapist to:
  * increase physical activity 30 minutes/day (At least 150 min/week) until 8 weeks postoperatively
  * decrease time spent sitting/lying
  The intervention includes a prescribed FaR (Fysisk aktivitet på recept) with frequency, duration and intensity of the activity corresponding 12-15 on the BORG-RPE scale.
  Arms: Increased physical activity
Other: Standard care
  Arms: Standard care

SUMMARY:
There are limited knowledge about the impact of increased pre-operative physical training on postoperative physical activity levels as well as on recovery and complication rates after bariatric surgery.

The primary aim of this study is to investigate whether an intervention including individual coaching to improve level of physical activity before and after gastric bypass surgery leads to a changed of level physical activity post-operatively at eight weeks, one and two years.

Secondary aims of the study are to investigate whether increased physical activity has effects on complication rates, re-admissions and re-operations, post-operative weight-loss, gastrointestinal pain, recovery measured as hospital stay, sick-leave and QoL, resumption of normal physical activity.

METHODS 300 patients will be recruited and randomized to an intervention group or control group. The patients in the intervention group will receive individual coaching by a physical therapist to:

* increase physical activity 30 minutes/day (At least 150 min/week)
* decrease time spent sitting/lying The patients in the control group will receive standard care.

Before surgery, 6 weeks, and one year after surgery patient will fill in a questionnaire including level of physical activity, sick leave, quality of life and gastrointestinal pain. In addition blood test will be taken and complication rates recorded.

ELIGIBILITY:
Inclusion Criterion:

- Patients at including hospitals scheduled for gastric bypass surgery

Exclusion Criteria:

* Inability to understand given information.
* Inability to perform the intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRES (IPAQ) | From inclusion 1 year postoperatively
  Physical activity level measured in METS (Metabolic Equivalent)
Saltin-Grimby Physical Activity Scale (SGPAS) | From inclusion to 1 year postoperatively
  Physical activity level, 1-4 (4 highest activity level).

SECONDARY OUTCOMES:
Complication rates | From inclusion to 30 days postoperatively
  Anastomotic leakages, bleedings that require intervention, thrombosis, re-admissions and re-operations derived from the patient medical records
Length of stay | From surgery to discharge. On average two days
  Days at hospital
Sick-leave | From surgery to at latest 1 year postoperatively
  Sick-leave is prescribed one week at a time, patients are required to call the doctor, to ask for prolonged sick-leave a week at a time.
Blood test- glucose metabolism | From surgery to 2 years postoperatively
  Glucose metabolism-
Blood test- Blood lipids | From surgery to 2 years postoperatively
  Metabolic change lipids
Blood tests, Blood sugar | From surgery to 2 years postoperatively
  HbA1c
Blood tests, fasting blood suger | From surgery to 2 years postoperatively
  Fasting P-glucose
Blood tests | From surgery to 2 years postoperatively
  Blood lipids
Weight | From surgery to 2 years postoperatively
  Actual weight measured during clinical visits
General Quality of Life, QoL By EQ5D | From inclusion 1 year postoperatively
  EQ5D, 5 questions with 3 different answers each (1 best value) leaving a 5 digit code which is transfered to a score from 0.3403-0.9694
Gastrointestinal pain by Gastrointestinal Symptom Rating Scale (GSRS) | From inclusion 1 year postoperatively
  Gastrointestinal Symptom Rating Scale, 16 questions rated on scales with 7 levels (a-low symptoms to g- worst symtoms)
Self reported co-morbidity | From inclusion 1 year postoperatively
  Number of patients with diabetes and with dyslipidemia medications
Self reported medication because of co-morbidity | From inclusion 1 year postoperatively
  Number of patients with medication because of diabetes, high blood pressure and dyslipidemia.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fagevik Olsén, pHd, Principal Investigator — Sahlgrenska Academy at Gothenburg university, Sweden
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schubert-Hjalmarsson E, Albertsson L, Englund E, Olsen MF. Joint Pain Outcomes After Metabolic and Bariatric Surgery in Patients With and Without Hypermobility. Obes Sci Pract. 2026 Jan 13;12(1):e70115. doi: 10.1002/osp4.70115. eCollection 2026 Feb. PMID 41541615